CLINICAL TRIAL: NCT00004159
Title: Biweekly Gemcitabine and Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer and Solid Tumors: A Phase I/IIa Study
Brief Title: Gemcitabine Plus Paclitaxel in Treating Patients With Advanced Non-small Cell Lung Cancer or Other Solid Tumor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067399; UAB-9720; UAB-F970730006; NCI-G99-1624
Record Dates: First submitted 1999-12-10; First posted 2004-07-26 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of gemcitabine plus paclitaxel in treating patients who have advanced non-small cell lung cancer or other solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicities of biweekly administration of gemcitabine and paclitaxel in patients with advanced non-small cell lung cancer (NSCLC) or other solid tumor. II. Determine the response rate, duration of response, and disease free interval for this patient population after this therapy.

OUTLINE: This is a dose escalation study. Patients receive paclitaxel IV over 1 hour followed 2 hours later by gemcitabine IV over 30 minutes on days 1, 15, and 29. Treatment repeats every 6 weeks for a maximum of 8 courses. Cohorts of 3-5 patients receive escalating doses of paclitaxel and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 patients experience dose limiting toxicity. Once the MTD is reached, an additional 14 patients (chemotherapy naive) with advanced NSCLC are treated at the recommended phase II dose. Patients are followed every 8 weeks for 6 months.

PROJECTED ACCRUAL: A minimum of 3 patients will be accrued for the phase I portion and a total of 14 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Phase I portion (closed for accrual after the maximum tolerated dose and dose limiting toxicity were determined) Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC) or other solid tumor for which no standard curative treatment exists Phase II portion (open for accrual): Histologically proven stage IV NSCLC without prior chemotherapy Measurable or evaluable disease No primary brain tumors Brain metastases allowed if controlled by radiation or stereotactic radiosurgery No lymphoproliferative disease No HIV related malignancies

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No congestive heart failure Other: Not pregnant or nursing Fertile patients must use effective contraception No serious nonmalignant disease No active/uncontrolled infection or bleeding (e.g., active peptic ulcer disease) No other primary malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix No allergy to Cremophor

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Phase I: No prior paclitaxel or gemcitabine At least 3 weeks since other prior chemotherapy and recovered Phase II: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-02; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, FACP, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States